CLINICAL TRIAL: NCT00170222
Title: The Value of Antibiotic Treatment of Exacerbations of Hospitalised COPD Patients
Brief Title: Placebo Versus Antibiotics in Acute Exacerbations of Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical Center Alkmaar (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M02-007
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Acute bronchitis; antibiotics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis | interventions — Doxycycline

INTERVENTIONS:
Drug: doxycycline

SUMMARY:
The role of antibiotic therapy in patients with COPD remains controversial. While the outcome of several clinical trials is in favour of antibiotics, the quality of these studies in insufficient. In this study the efficacy of doxycycline is compared to placebo. All concommitant treatment (steroids, bronchodilator therapy, physiotherapy) is standardized.

The investigators hypothesize that patients with an acute exacerbations will have a better outcome when treated with antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Acute exacerbation of COPD type I or II according to GOLD
* Ability to perform lung function tests
* Ability to take oral medication

Exclusion Criteria:

* Pregnant or lactating women, or women of childbearing age not using an acceptable method of contraception.
* Pretreatment ( > 24 hours) with an antibiotic for the present exacerbation.
* Pretreatment with corticosteroids (>30 mg for more than 4 days) for the present exacerbation.
* Progression or new radiographic abnormalities on the chest X-ray.
* Severe exacerbation that required mechanical ventilation.
* History of bronchiectasis
* Recent or unresolved lung malignancy.
* Other disease likely to require antibiotic therapy.
* Significant gastrointestinal or other conditions that may affect study drug absorption.
* Class III or IV congestive heart failure or stroke.
* Immunodeficiency disorders such as AIDS, humoral immune defect, ciliary dysfunction etc. and the use of immunosuppressive drugs (>30 mg prednisolone maintenance dose or equivalent for more than 4 weeks).
* Cystic fibrosis
* Tuberculosis.
* Impaired renal function (creatinine clearance < 20 ml/min).

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2002-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy at the end of treatment

SECONDARY OUTCOMES:
Treatment failure at follow up
Number of exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Johannes MA Daniels, drs, Principal Investigator — Pulmo Science; Dominic Snijders, drs, Principal Investigator — Pulmo Science
Locations (1):
- Medisch centrum Alkmaar, Alkmaar, North Holland, Netherlands

REFERENCES:
- [Derived] Daniels JM, Schoorl M, Snijders D, Knol DL, Lutter R, Jansen HM, Boersma WG. Procalcitonin vs C-reactive protein as predictive markers of response to antibiotic therapy in acute exacerbations of COPD. Chest. 2010 Nov;138(5):1108-15. doi: 10.1378/chest.09-2927. Epub 2010 Jun 24. PMID 20576731
- [Derived] Daniels JM, Snijders D, de Graaff CS, Vlaspolder F, Jansen HM, Boersma WG. Antibiotics in addition to systemic corticosteroids for acute exacerbations of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2010 Jan 15;181(2):150-7. doi: 10.1164/rccm.200906-0837OC. Epub 2009 Oct 29. PMID 19875685